CLINICAL TRIAL: NCT00287703
Title: Pulsed Electro Magnetic Fields (PEMF) Treatment in Patients With Treatment-Resistant Major Depression in Ongoing Pharmacological Treatment of Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: The Lundbeckfoundation (Unknown); Biofields (Unknown)
Responsible Party: Klaus Martiny, Psychiatric Research Unit, Hillerod Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Final version 26 Oktober 2005
Record Dates: First submitted 2006-01-31; First posted 2006-02-07 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Depression
Keywords: Major depression; Treatment resistant; PEMF; AQT; Hamilton
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active Pulsating Electro Magnetic Fields (PEMF) treatment
  Interventions: Device: Pulsating Electro-Magnetic Fields
- 2 (Sham Comparator): 5 days a week for 5 weeks for 30 minutes Sham PEMF
  Interventions: Device: Pulsating Electro-Magnetic Fields sham

INTERVENTIONS:
Device: Pulsating Electro-Magnetic Fields — 5 days a week for 5 weeks 30 minutes
  Arms: 1
Device: Pulsating Electro-Magnetic Fields sham — sham PEMF
  Arms: 2

SUMMARY:
About 30% of patients with major depression are treatment resistant to pharmacological treatment. In the search for new methods to treat depression a great interest has been put into the use of electromagnetic fields. This study tests the hypothesis that ultra-weak electromagnetic fields with a specific wave pattern (PEMF = pulsed electro magnetic fields) can alleviate the symptoms of depression.

DETAILED DESCRIPTION:
In this study, a patient with treatment resistant depression, as defined by Harold Sackeim, is subjected to 5 weeks of treatment with active or sham PEMF treatment for 30 minutes on every working day. The pharmacological treatment for depression is maintained unaltered throughout the study. Depression severity is measured at the beginning of the study and at each weekly visit. Side effects are closely observed. The ability to concentrate is measured by the AQT test (Alzheimers Quick Test). Personality is assessed by use of the SCID-II-instrument (DSM-IV axis II).

ELIGIBILITY:
Inclusion Criteria:

* Major depression
* Treatment resistance
* Age above 18 years
* Hamilton 17 item score above 13
* Unaltered pharmacological treatment in last 4 weeks

Exclusion Criteria:

* Psychotic disorder
* Mental retardation
* Suicidality
* Earlier treatment with PEMF
* Abuse of alcohol or other substances
* Patient not able to come to appointed visits
* Antisocial, borderline or schizotypic personality disorder
* Women lactating or pregnant
* Unreliable contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale score (depression) | 1 week

SECONDARY OUTCOMES:
AQT, measure of concentration | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Martiny, MD, Ph.D., Principal Investigator — Psychiatric Research Unit Fredericksburg General Hospital
Locations (1):
- Speciallægerne Falkoner Allé, Municipality of Frederiksberg, Denmark

REFERENCES:
- [Derived] Martiny K, Lunde M, Bech P. Transcranial low voltage pulsed electromagnetic fields in patients with treatment-resistant depression. Biol Psychiatry. 2010 Jul 15;68(2):163-9. doi: 10.1016/j.biopsych.2010.02.017. Epub 2010 Apr 10. PMID 20385376